CLINICAL TRIAL: NCT07127042
Title: A Randomized, Double-blind, Active-controlled, Multicenter Clinical Study to Evaluate the Efficacy and Safety of BT-114143 Injection in Reducing Perioperative Blood Loss in Unilateral Total Knee Arthroplasty
Brief Title: Study on BT-114143 Reducing Perioperative Bleeding in Total Knee Arthroplasty（TKA）
Acronym: TKA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ScinnoHub Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-114143-II-01
Record Dates: First submitted 2025-07-18; First posted 2025-08-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose Group (Experimental): High-dose BT-114143
  Interventions: Drug: High-dose BT-14143
- Low-dose Group (Experimental): Low-dose BT-114143
  Interventions: Drug: Low-dose BT-114143
- Control Group (Active Comparator): Tranexamic acid
  Interventions: Drug: Tranexamic Acid (IV)

INTERVENTIONS:
Drug: Low-dose BT-114143 — Intravenous infusion of BT-114143 Injection is started 10-15 minutes before skin incision at a Low-dose BT-114143, and 50mL of normal saline is administered intravenously 3 hours (±10 minutes) after the end of the surgery.
  Arms: Low-dose Group
Drug: High-dose BT-14143 — Intravenous infusion of BT-114143 Injection is started 10-15 minutes before skin incision at a High-dose BT-114143, and 50mL of normal saline is administered intravenously 3 hours (±10 minutes) after the end of the surgery.
  Arms: High-dose Group
Drug: Tranexamic Acid (IV) — Intravenous infusion of TXA is started 10-15 minutes before skin incision at a dose of 20mg/kg, and intravenous infusion of TXA is initiated 3 hours (±10 minutes) after the end of the surgery at a dose of 1g.
  Arms: Control Group

SUMMARY:
This is a randomized, double-blind, active-controlled, multicenter, phase II clinical study designed to evaluate the efficacy and safety of BT-114143 Injection in the perioperative treatment of unilateral total knee arthroplasty. It is planned to enroll 270 subjects undergoing elective unilateral open total knee arthroplasty. Subjects will be randomly assigned to the BT-114143 high-dose group, BT-114143 low-dose group, or tranexamic acid treatment group in a 1:1:1 ratio. All subjects will receive intravenous injection of BT-114143 or tranexamic acid before and after surgical incision. The total perioperative blood loss in different treatment groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years, regardless of gender (including boundary values);
* Patients with osteoarthritis who meet the diagnostic criteria of the American College of Rheumatology (ACR), meet the indications for knee replacement, and plan to undergo total knee arthroplasty;
* American Society of Anesthesiologists (ASA) physical status classification ≤ Grade 3;
* Patients with mild knee deformity: flexion deformity < 20°, varus deformity < 15°-5.No abnormalities in preoperative platelet level and coagulation function;
* Body Mass Index [BMI = weight (kg)/height² (m²)] within the range of 20.0-35.0 kg/m² (including critical values);
* Patients voluntarily sign the informed consent form.

Exclusion Criteria:

* Uncontrolled systemic or local infections, including but not limited to pulmonary infection, skin infection, urinary tract infection, etc.;
* Serum albumin concentration < 35g/L;
* Patients with preoperative hemoglobin < 110g/L;
* Patients with a known history of severe venous thromboembolism or those with severe thromboembolic risk indicated by lower extremity venous ultrasound (such as popliteal vein and proximal venous thrombosis);
* Patients with severe cardiovascular and cerebrovascular diseases (history of myocardial infarction, angina pectoris, stroke, epileptic seizure, subarachnoid hemorrhage, heart failure, etc. within 6 months before screening);
* Patients with severe varicose veins or severe peripheral arterial diseases affecting distal blood supply (lower extremity arterial stenosis, occlusion);
* Patients with cancer within 5 years before screening, except for cured skin basal cell carcinoma;
* Hypertensive patients with poorly controlled blood pressure (SBP ≥ 140mmHg and/or DBP ≥ 90mmHg), or those requiring combined use of thiazide diuretics, loop diuretics, potassium-sparing diuretics, etc;
* Patients with poorly controlled diabetes (fasting blood glucose > 8 mmol/L);
* Patients with known severe history of allergic reactions that may affect the evaluation of the study, or those allergic to tranexamic acid and its similar drugs;
* Patients who have undergone open knee surgery on the ipsilateral knee (arthroscopic surgery is allowed);
* Patients planning to undergo other surgeries within 1 month (including simultaneous bilateral total knee arthroplasty);
* Patients with combined severe liver or kidney dysfunction (eGFR < 60 mL/min/1.73 m², ALT and/or AST > 2 times the upper limit of normal range);
* Positive for hepatitis B surface antigen, hepatitis C antibody, HIV antigen/antibody, or syphilis antibody during screening;
* Patients who have used drugs affecting coagulation function within 1 week before surgery (such as aspirin, clopidogrel, ticlopidine, dipyridamole, ginkgo biloba preparations, heparin, warfarin, citrate, hemocoagulase, vitamin K, antifibrinolytic agents, etamsylate, etc.);
* Patients who have used drugs with risks of bleeding and thrombosis within 1 week before surgery, such as oral contraceptives, estrogens, or prothrombin complex concentrates;
* Patients who have used drugs that can increase hemoglobin levels (such as erythropoietin, EPO) within 4 weeks before screening;
* 1-Patients who have taken iron supplements within 1 week before surgery or used intravenous iron supplements within 4 weeks before surgery.
* Patients with mental or neurological diseases, a history of drug abuse, or a history of alcoholism that, in the investigator's opinion, could affect their -participation in the study,specifically, those who consumed more than 14 standard units of alcohol per week within 3 months before screening (1 standard unit equals 14g of alcohol, such as 360ml of beer, 45ml of spirits with 40% alcohol content, or 150ml of wine);
* Patients who have participated in or are currently participating in other clinical trials within 3 months before screening (participation in a clinical trial is defined as the patient receiving an intervention);
* Pregnant or lactating women, or patients of childbearing potential who cannot ensure the use of at least one acceptable form of contraception during the study and for 3 months after the end of the study;
* Patients whom the investigator deems unsuitable for participation in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total blood loss | The 3rd day after surgery
  The blood loss was calculated using the Gross formula based on changes in hematocrit (HCT) from the subjects' preoperative and postoperative blood routine tests.

SECONDARY OUTCOMES:
Occult blood loss | The 3rd day after surgery
  Occult blood loss = Total blood loss - Intraoperative blood loss (no drainage tube is placed postoperatively)
Total blood loss on the first day after surgery | The first day after surgery
  The blood loss was calculated using the Gross formula based on changes in hematocrit (HCT) from the subjects' preoperative and postoperative blood routine tests.
Allogeneic blood transfusion rate | The 3rd day after surgery
Allogeneic blood transfusion volume | The 3rd day after surgery
Changes in hemoglobin levels from baseline | The 3rd day after surgery
Changes in hematocrit levels from baseline | The 3rd day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics, West China Hospital, SIchuan University, Chengdu, Si'Chuan, China

IPD SHARING:
Plan to Share IPD: No